CLINICAL TRIAL: NCT02647580
Title: Appetite-regulating Hormones, the Gut Microbiome and the Metabolome in Children With Failure to Thrive
Brief Title: Appetite Regulation in Children With Failure to Thrive
Status: Completed | Type: Observational
Sponsor: Lena Kirchner Brahe (Other)
Collaborators: Hvidovre University Hospital (Other); Technical University of Denmark (Other)
Responsible Party: Sponsor-Investigator, Lena Kirchner Brahe, Assistant professor, PhD, University of Copenhagen
Organization: University of Copenhagen (Other)
Other Study IDs: M229
Record Dates: First submitted 2015-12-21; First posted 2016-01-06 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Failure to Thrive
Keywords: Growth; Children; Appetite-regulating hormones; Gut Microbiota
MeSH Terms: conditions — Failure to Thrive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma, serum, feces, urine
Oversight: Data Monitoring Committee: No

SUMMARY:
Failure to thrive (FTT) is an expression for inadequate growth in the early childhood and thus, a sign of undernutrition. This study will include children with FTT, and compare with existing data from children with normal and excessive growth.

The overall aim of this study is to explore whether 1) children who develop FTT with no organic explanation differ from healthy normal weight and overweight children in their basal level of appetite-regulating hormones and 2) if inadequate, normal and excessive growth in children can be partly predicted by variation in their gut microbiome and metabolome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with failure to thrive
* Weight for height > 1.9 SD below the median by use of the WHO Child Growth Standards
* Age between 12-36 months

Exclusion Criteria:

* Cancer
* Inflammatory bowel disease
* Celiac disease
* Immunodeficiency
* Other somatic disease that can explain the growth failure

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with failure to thrive
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Appetite-regulating hormones (ghrelin, PYY, leptin) measured by fasting blood samples | At subject enrollment

SECONDARY OUTCOMES:
Microbiota composition measured by fecal samples | At subject enrollment
Metabolome measured by urine samples | At subject enrollment
Metabolic markers (insulin, glucose) measured by fasting blood samples | At subject enrollment
Body weight measured in kilograms | At subject enrollment
Height measured in centimeters | At subject enrollment
Head circumference measured in centimeters | At subject enrollment
Waist circumference measured in centimeters | At subject enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark